CLINICAL TRIAL: NCT05663788
Title: Web-based Learning Module to Increase the Accuracy of Optical Diagnosis for Detecting the Invasive Pattern of Colorectal Polyps (LODIP Study). Randomised Controlled Trial
Brief Title: Web-based Learning Module on Optical Diagnosis of Early Colorectal Cancer
Acronym: LODIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Althaia Xarxa Assistencial Universitària de Manresa (Other)
Collaborators: Fundació La Marató de TV3 (Other); Spanish Society of Digestive Endoscopy (Other); Asociación Española de Gastroenterología (Other)
Responsible Party: Principal Investigator, Ignasi Puig, Gastroenterology Consultant, Principal Investigator, Althaia Xarxa Assistencial Universitària de Manresa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CEI 19/18
Record Dates: First submitted 2022-12-07; First posted 2022-12-23 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer; Colorectal Cancer Stage I
Keywords: advance endoscopy; collaborative research; colonoscopy; early colorectal cancer; colorectal polyps; optical diagnosis; training; invasive pattern; magnifying endoscopy; chromoendoscopy; deep submucosal invasion
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Non-pharmacological multi-centre, stratified (by the centre and experience, with balance randomisation [1:1]), randomised, controlled, parallel trial conducted in Spain.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-learning module gastroenterologists (Experimental): Gastroenterologists participating in the e-learning module
  Interventions: Other: E-learning module
- Control group (No Intervention): Gastroenterologists not participating in the e-learning module

INTERVENTIONS:
Other: E-learning module — The intervention is a structured e-learning module on a web-based platform (www.trainingopticaldiagnosis.com) that consists of:
  * 10 modules, including theoretical knowledge and multiple exercises.
  * 2 seminars with a tutor (after Module 5 and Module 10)
  * feedback from the tutor on three cases recorded by the participant.
  * 20-images test before and after the content described above (10 Modules, 2 seminars with tutors and feedback on three cases)
  All the Gastroenterologists participating in the study will predict deep submucosal invasion in their routine colonoscopies and will register clinical outcomes during 12 months. The randomisation and intervention will be conducted 6 months after starting to predict deep submucosal invasion and registering clinical outcomes.
  Arms: E-learning module gastroenterologists

SUMMARY:
International guidelines recommend deciding the treatment of colorectal lesions based on the estimated histology by endoscopic optical diagnosis. However, the theoretical and practical knowledge on optical diagnosis is not widely expanded

The mail goal of this randomised controlled trial is to compare the pooled sensitivity of optical diagnosis for predicting deep submucosal invasion in large non-pedunculated polyps > 20 mm assessed in routine colonoscopies of gastroenterologists attending a e-learning module (intervention group) vs gastroenterologists who do not (control group)

The main questions the study aims to answer are:

* Is the pooled sensitivity of optical diagnosis for predicting deep submucosal invasion in large non-pedunculated polyps assessed in routine colonoscopies increased in those gastroenterologists participating in the e-learning module?
* Is the pooled diagnostic accuracy of optical diagnosis for predicting deep sm invasion in large non-pedunculated polyps ≥ 20 mm assessed in routine colonoscopies increased in those gastroenterologists participating in the e-learning module?
* In lesions with submucosal invasion, is the en bloc and complete resection rate (R0) increased in those gastroenterologists participating in the e-learning module?
* In lesions referred to surgery, is the pooled benign polyps rate decreased in those gastroenterologists participating in the e-learning module?
* In lesions treated with advanced en bloc procedures (ESD, TAMIS, fullthickness resection), is the pooled rate of histology with high-grade dysplasia, intramucosal cancer or submucosal invasion increased in those gastroenterologists participating in the e-learning module?
* In lesions treated with piecemeal endoscopic resection, is the pooled rate of histology with high-grade dysplasia, intramucosal cancer or submucosal invasion decreased in those gastroenterologists participating in the e-learning module?
* Is the diagnostic accuracy for predicting deep submucosal invasion in a test with pictures increased after participating in the e-learning module?

The participants (or subjects of study) are gastroenterologists. They will be randomised to do the e-learning course (intervention group) or not (control group).

Researchers will compare clinical outcomes of gastroenterologists participating in the e-learning module vs gastroenterologists not participating in the e-learning module to see if:

* the pooled sensitivity of optical diagnosis for predicting deep submucosal invasion in large non-pedunculated polyps > 20 mm assessed in routine colonoscopies is increased.
* the pooled diagnostic accuracy of optical diagnosis for predicting deep sm invasion in large non-pedunculated polyps > 20 mm is increased.
* the en bloc and complete resection rate (R0) is increased in lesions with submucosal invasion.
* the pooled benign polyps rate decreased in lesions referred to surgery.
* the pooled rate of histology with high-grade dysplasia, intramucosal cancer or submucosal invasion increased in lesions treated with advanced en bloc procedures (ESD, TAMIS, fullthickness resection).
* the pooled rate of histology with high-grade dysplasia, intramucosal cancer or submucosal invasion decreased in lesions treated with piecemeal endoscopic resection.
* the diagnostic accuracy for predicting deep submucosal invasion in a test with pictures after participating is increased.

DETAILED DESCRIPTION:
Non-pharmacological multi-centre randomised controlled trial. Gastroenterologists who have performed > 300 colonoscopies without supervision and who have finished/will finish the residency in Gastroenterology between 2014 and 2023 will be invited to participate. Gastroenterologists participating in the study will register the optical diagnosis, endoscopic lesions' characteristics, histology and clinical outcomes of consecutive non-pedunculated lesions ≥ 20 mm found in routine colonoscopies during a whole year. Participants allocated in the intervention group will receive a learning module after six months. Those assigned in the control group will not receive any learning module (they will be offered to do it at the end of the study). Pooled sensitivity and diagnostic accuracy of optical diagnosis for predicting deep submucosal invasion, and clinical outcomes in routine colonoscopies will be compared in both groups. Diagnostic accuracy for predicting deep submucosal invasion in a test with pictures before and after participating will also be compared.

ELIGIBILITY:
Inclusion Criteria:

* Gastroenterologists who have performed > 300 colonoscopies without supervision and are in the last training year or had finished the Gastroenterology residency after 2014.

Exclusion Criteria:

* Endoscopists who have learned the invasive pattern in a centre where endoscopists have published a high diagnostic accuracy for predicting deep submucosal invasion (Japanese centres).

Min Age: 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Pooled sensitivity of endoscopic optical diagnosis for predicting deep submucosal invasion in routine colonoscopies | immediately after the colonoscopy
  Pooled sensitivity of endoscopic optical diagnosis (test assessed by Gastroenterologists according to the ESGE guidelines) for predicting deep submucosal invasion (gold standard measured by the Pathologists according to the WHO criteria) in routine colonoscopies.

SECONDARY OUTCOMES:
Pooled Sensitivity of endoscopic optical diagnosis for predicting deep submucosal invasion | immediately after the colonoscopy
  Pooled Sensitivity of endoscopic optical diagnosis (test assessed by Gastroenterologists according to the ESGE guidelines) for predicting deep submucosal invasion (gold standard measured by the Pathologists according to the WHO criteria) in routine colonoscopies.
Pooled Specificity of endoscopic optical diagnosis for predicting deep submucosal invasion | immediately after the colonoscopy
  Pooled Specificity of endoscopic optical diagnosis (test assessed by Gastroenterologists according to the ESGE guidelines) for predicting deep submucosal invasion (gold standard measured by the Pathologists according to the WHO criteria) in routine colonoscopies.
Pooled ROC area of endoscopic optical diagnosis for predicting deep submucosal invasion | immediately after the colonoscopy
  Pooled ROC area of endoscopic optical diagnosis (test assessed by Gastroenterologists according to the ESGE guidelines) for predicting deep submucosal invasion (gold standard measured by the Pathologists according to the WHO criteria) in routine colonoscopies.
Pooled PPV of endoscopic optical diagnosis for predicting deep submucosal invasion | immediately after the colonoscopy
  Pooled PPV of endoscopic optical diagnosis (test assessed by Gastroenterologists according to the ESGE guidelines) for predicting deep submucosal invasion (gold standard measured by the Pathologists according to the WHO criteria) in routine colonoscopies.
Pooled NPV of endoscopic optical diagnosis for predicting deep submucosal invasion | immediately after the colonoscopy
  Pooled NPV of endoscopic optical diagnosis (test assessed by Gastroenterologists according to the ESGE guidelines) for predicting deep submucosal invasion (gold standard measured by the Pathologists according to the WHO criteria) in routine colonoscopies.
Pooled LR+ of endoscopic optical diagnosis for predicting deep submucosal invasion | immediately after the colonoscopy
  Pooled LR+ of endoscopic optical diagnosis (test assessed by Gastroenterologists according to the ESGE guidelines) for predicting deep submucosal invasion (gold standard measured by the Pathologists according to the WHO criteria) in routine colonoscopies.
Pooled LR- of endoscopic optical diagnosis for predicting deep submucosal invasion | immediately after the colonoscopy
  Pooled LR- of endoscopic optical diagnosis (test assessed by Gastroenterologists according to the ESGE guidelines) for predicting deep submucosal invasion (gold standard measured by the Pathologists according to the WHO criteria) in routine colonoscopies.
Pooled en bloc resection rate in polyps containing submucosal invasion | immediately after the colonoscopy
  Pooled en bloc resection rate in polyps containing submucosal invasion found in routine colonoscopies
Pooled complete resection rate (R0) in polyps containing submucosal invasion | immediately after the colonoscopy
  Pooled complete resection rate (R0) according to the pathologist criteria in polyps containing submucosal invasion
Pooled benign polyps rate in lesions refered to surgery | immediately after the colonoscopy
  Pooled benign polyps rate in lesions refered to surgery
Pooled rate of histology with high-grade dysplasia, intramucosal cancer or submucosal invasion in lesions treated with advanced en bloc procedures (ESD, TAMIS, fullthickness resection) | immediately after the colonoscopy
  Pooled rate of histology with high-grade dysplasia, intramucosal cancer or submucosal invasion in lesions treated with advanced en bloc procedures (ESD, TAMIS, fullthickness resection)
Pooled rate of histology with high-grade dysplasia, intramucosal cancer or submucosal invasion in lesions treated with piecemeal endoscopic resection | immediately after the colonoscopy
  Pooled rate of histology with high-grade dysplasia, intramucosal cancer or submucosal invasion in lesions treated with piecemeal endoscopic resection
Pooled Sensitivity of endoscopic optical diagnosis for predicting deep submucosal invasion in a 20-image test before and after the learning module in the intervention group | immediately after the colonoscopy
  Pooled Sensitivity of endoscopic optical diagnosis for predicting deep submucosal invasion in a 20-image test before and after the learning module in the intervention group
Pooled Specificity of endoscopic optical diagnosis for predicting deep submucosal invasion in a 20-image test before and after the learning module in the intervention group | immediately after the colonoscopy
  Pooled Specificity of endoscopic optical diagnosis for predicting deep submucosal invasion in a 20-image test before and after the learning module in the intervention group
Pooled ROC area of endoscopic optical diagnosis for predicting deep submucosal invasion in a 20-image test before and after the learning module in the intervention group | immediately after the colonoscopy
  Pooled ROC area of endoscopic optical diagnosis for predicting deep submucosal invasion in a 20-image test before and after the learning module in the intervention group
Pooled PPV of endoscopic optical diagnosis for predicting deep submucosal invasion in a 20-image test before and after the learning module in the intervention group | immediately after the colonoscopy
  Pooled PPV of endoscopic optical diagnosis for predicting deep submucosal invasion in a 20-image test before and after the learning module in the intervention group
Pooled NPV of endoscopic optical diagnosis for predicting deep submucosal invasion in a 20-image test before and after the learning module in the intervention group | immediately after the colonoscopy
  Pooled NPV of endoscopic optical diagnosis for predicting deep submucosal invasion in a 20-image test before and after the learning module in the intervention group
Pooled LR+ of endoscopic optical diagnosis for predicting deep submucosal invasion in a 20-image test before and after the learning module in the intervention group | immediately after the colonoscopy
  Pooled LR+ of endoscopic optical diagnosis for predicting deep submucosal invasion in a 20-image test before and after the learning module in the intervention group
Pooled LR- of endoscopic optical diagnosis for predicting deep submucosal invasion in a 20-image test before and after the learning module in the intervention group | immediately after the colonoscopy
  Pooled LR- of endoscopic optical diagnosis for predicting deep submucosal invasion in a 20-image test before and after the learning module in the intervention group

CONTACTS AND LOCATIONS:
Overall Officials: Ignasi Puig, PhD, Principal Investigator — Althaia Xarxa Assistencial Universitària de Manresa
Locations (12):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States
- National Cancer Center, Chūō, Tokyo, Japan
- Spain (9):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Althaia Xarxa Assistencial Universitària de Manresa, Manresa, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Comarcal de Alcañiz, Alcañiz, Teruel
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitari i Politècnic La Fe, Valencia
- Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Puig I, Lopez-Ceron M, Arnau A, Rosinol O, Cuatrecasas M, Herreros-de-Tejada A, Ferrandez A, Serra-Burriel M, Nogales O, Vida F, de Castro L, Lopez-Vicente J, Vega P, Alvarez-Gonzalez MA, Gonzalez-Santiago J, Hernandez-Conde M, Diez-Redondo P, Rivero-Sanchez L, Gimeno-Garcia AZ, Burgos A, Garcia-Alonso FJ, Bustamante-Balen M, Martinez-Bauer E, Penas B, Pellise M; EndoCAR group, Spanish Gastroenterological Association and the Spanish Digestive Endoscopy Society. Accuracy of the Narrow-Band Imaging International Colorectal Endoscopic Classification System in Identification of Deep Invasion in Colorectal Polyps. Gastroenterology. 2019 Jan;156(1):75-87. doi: 10.1053/j.gastro.2018.10.004. Epub 2018 Oct 6. PMID 30296432
- [Background] Bisschops R, East JE, Hassan C, Hazewinkel Y, Kaminski MF, Neumann H, Pellise M, Antonelli G, Bustamante Balen M, Coron E, Cortas G, Iacucci M, Yuichi M, Longcroft-Wheaton G, Mouzyka S, Pilonis N, Puig I, van Hooft JE, Dekker E. Advanced imaging for detection and differentiation of colorectal neoplasia: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2019. Endoscopy. 2019 Dec;51(12):1155-1179. doi: 10.1055/a-1031-7657. Epub 2019 Nov 11. PMID 31711241
- [Background] Kaminski MF, Hassan C, Bisschops R, Pohl J, Pellise M, Dekker E, Ignjatovic-Wilson A, Hoffman A, Longcroft-Wheaton G, Heresbach D, Dumonceau JM, East JE. Advanced imaging for detection and differentiation of colorectal neoplasia: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2014 May;46(5):435-49. doi: 10.1055/s-0034-1365348. Epub 2014 Mar 17. PMID 24639382
- [Background] Dekker E, Houwen BBSL, Puig I, Bustamante-Balen M, Coron E, Dobru DE, Kuvaev R, Neumann H, Johnson G, Pimentel-Nunes P, Sanders DS, Dinis-Ribeiro M, Arvanitakis M, Ponchon T, East JE, Bisschops R. Curriculum for optical diagnosis training in Europe: European Society of Gastrointestinal Endoscopy (ESGE) Position Statement. Endoscopy. 2020 Oct;52(10):899-923. doi: 10.1055/a-1231-5123. Epub 2020 Sep 3. PMID 32882737
- See also: website of the research group holding the e-learning platform — http://goesresearchgroup.com